CLINICAL TRIAL: NCT02322099
Title: A Multi-centre, Prospective, Randomised Trial of Short Course Alendronate Therapy or Placebo Combined With Vitamin D and Calcium to Prevent Loss of Bone Mineral Density in Antiretroviral-naïve, HIV-1 Infected Subjects Initiating Antiretroviral Therapy
Brief Title: Alendronate for Prevention of AntiRetroviral Therapy-associated Bone Loss
Acronym: APART
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Due to the COVID-19 pandemic the study was terminated prematurely
Sponsor: University College Dublin (Other)
Collaborators: Health Research Board, Ireland (Other); Royal College of Surgeons, Ireland (Other); Mater Misericordiae University Hospital (Other); Beaumont Hospital (Other); Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Patrick Mallon, Principal Investigator, University College Dublin
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: APART_2014
Record Dates: First submitted 2014-12-17; First posted 2014-12-22 (Estimated); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Bone Demineralization
Keywords: human immunodeficiency virus; bone diseases; osteopenia; osteoporosis; fracture; bone turnover; alendronate; antiretroviral
MeSH Terms: conditions — Bone Demineralization, Pathologic; Acquired Immunodeficiency Syndrome; Bone Diseases; Bone Diseases, Metabolic; Osteoporosis; Fractures, Bone | interventions — Alendronate; Calcium Carbonate; Cholecalciferol; Tenofovir; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Alendronate (Active Comparator): Alendronate 70 mg plus calcium/vitamin D (1250 mg/400iu) plus Truvada®
  Interventions: Drug: Alendronate; Dietary Supplement: calcium carbonate and colecalciferol; Drug: Tenofovir disoproxil
- Placebo (Placebo Comparator): Placebo to alendronate 70mg plus calcium/vitamin D (1250 mg/400iu) plus Truvada®
  Interventions: Drug: Placebo; Dietary Supplement: calcium carbonate and colecalciferol; Drug: Tenofovir disoproxil

INTERVENTIONS:
Drug: Alendronate — alendronate 70 mg tablets to be administered weekly for a total of 14 weeks, commencing 2 weeks prior to ART initiation
  Other Names: Fosamax; Romax
  Arms: Alendronate
Drug: Placebo — Sugar pill manufactured to mimic alendronate 70 mg tablet administered weekly for a total of 14 weeks, commencing 2 weeks prior to ART
  Arms: Placebo
Dietary Supplement: calcium carbonate and colecalciferol — Calcium carbonate 1250 mg (equivalent to 500 mg of elemental calcium) and colecalciferol 400 iu (equivalent to 10 micrograms of vitamin D3) tablets administered twice daily for a total of 14 weeks, commencing 2 weeks prior to ART initiation
  Other Names: Calcichew D3 forte; Ideos
Drug: Tenofovir disoproxil — Emtricitabine / tenofovir disoproxil fumarate 200 / 300 mg tablet administered once-daily with food (open-label) commencing 2 weeks after alendronate initiation and continuing for 48 weeks
  Other Names: Truvada

SUMMARY:
Antiretroviral therapy (ART) initiation is associated with a significant loss of bone mineral density (BMD), characterised by increases in bone turnover, which is largely limited to the first 48 weeks of therapy. Bisphosphonates, such as alendronate, decrease bone turnover and can limit loss of bone mineral density.

This study aims to determine if a short course of treatment with the oral bisphosphonate alendronate can limit loss of bone mineral density associated with initiation of ART in HIV-1 infected, antiretroviral naive, adult subjects.

DETAILED DESCRIPTION:
Multi-centre, prospective, randomised, double-blind, placebo-controlled trial over 50 weeks. The aims of this study include:

1. To determine if short-course treatment with alendronate versus placebo combined with calcium and vitamin D, initiated 2 weeks prior to start of ART and can prevent loss of BMD over 48 weeks of follow-up post ART initiation.
2. To explore the effect of alendronate on bone turnover in the setting of ART initiation.
3. To determine which factors, such as choice of ART, impacts the protective effect of alendronate in preventing BMD loss.
4. To determine the relationship between changes in bone turnover markers, vitamin D, parathyroid hormone and calcium levels.
5. To explore the pathogenesis of BMD loss with initiation of ART by investigating relationships between changes in immune function (T-cells and B-cells subsets), bone turnover and BMD.

ELIGIBILITY:
Inclusion Criteria:

* male>30 years old or female>35 years old
* HIV-1 antibody positive
* antiretroviral therapy naïve
* be presumed to have achieved peak bone mass
* be eligible for initiation of antiretroviral therapy in the opinion of the investigator
* be able to provide written, informed consent

Exclusion Criteria:

* subjects unable to comply with the study protocol or unable to stand/sit upright for at least 30 minutes
* history of osteoporosis
* history of fragility fracture or previous femoral fracture
* chronic renal failure
* hypocalcemia or hypercalcemia at screening
* history of Paget's disease or known primary hyperparathyroidism
* previous treatment with or allergy (including hypersensitivity) to bisphosphonates
* recent history (past 12 months) of peptic or duodenal ulcers or oesophagitis, aspiration or any other abnormality of the oesophagus
* current therapy with prescribed calcium or vitamin D preparations (other than over-the-counter multivitamin preparations)
* current therapy with aspirin or other regularly prescribed non-steroidal anti-inflammatory drugs
* recent dental work (within the past 3 months) or poor oral hygiene (as judged in the opinion of the investigator)
* recent (within the past three months) significant steroid exposure
* for female subjects: pregnancy at screening, planning future pregnancies or unwilling to take measures to avoid pregnancy for the duration of the study
* where in the investigator's opinion, there is a necessity to initiate ART within the pre-ART study window period
* hepatitis B or hepatitis C co-infection
* any active illness (including AIDS illness) which in the opinion of the investigator precludes participation in the study
* subjects concurrently enrolled in another clinical trial of an investigational medical product

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2016-05; Primary Completion 2019-09 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Rate of changes in bone mineral density | 50 weeks
  Between-group differences in percentage change in total hip, lumbar spine, femoral neck BMD and body composition to week 50 among subjects who received at least one dose of the study medication

SECONDARY OUTCOMES:
Rate of changes in bone turnover markers | 50 weeks
  Between-group differences in percentage change in bone turnover markers
Impact of ART choice on alendronate protective effect | 50 weeks
  Impact of choice of ART on changes in BMD and bone turnover markers

OTHER OUTCOMES:
Pathogenesis of BMD loss with initiation of ART | 50 weeks
  Relationship between changes in T-cell and B-cell subsets, bone turnover and BMD with ART initiation

CONTACTS AND LOCATIONS:
Overall Officials: Patrick WG Mallon, MB BCh BAO,PhD,FRCPI, Principal Investigator — University College Dublin
Locations (2):
- Ireland (2):
  - Mater Misericordiae University Hospital, Dublin
  - Beaumont Hospital, Dublin

REFERENCES:
- [Background] Cotter AG, Sabin CA, Simelane S, Macken A, Kavanagh E, Brady JJ, McCarthy G, Compston J, Mallon PW; HIV UPBEAT Study Group. Relative contribution of HIV infection, demographics and body mass index to bone mineral density. AIDS. 2014 Sep 10;28(14):2051-60. doi: 10.1097/QAD.0000000000000353. PMID 25265073
- [Background] McComsey GA, Kendall MA, Tebas P, Swindells S, Hogg E, Alston-Smith B, Suckow C, Gopalakrishnan G, Benson C, Wohl DA. Alendronate with calcium and vitamin D supplementation is safe and effective for the treatment of decreased bone mineral density in HIV. AIDS. 2007 Nov 30;21(18):2473-82. doi: 10.1097/QAD.0b013e3282ef961d. PMID 18025884